CLINICAL TRIAL: NCT06037590
Title: A Pilot Open-label, Randomized, Crossover, Comparative Bioavailability Study of Levodopa Administered Via Levodopa Cyclops® (Test Product) Relative to INBRIJA® (Reference Product) in Healthy Adult Subjects
Brief Title: A Pilot Comparative Bioavailability Study of Levodopa Administered Via Levodopa Cyclops® Relative to INBRIJA®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PureIMS B.V. (Industry)
Collaborators: Cooperative Clinical Drug Research and Development AG (CCDRD AG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-504687-42-00
Record Dates: First submitted 2023-08-24; First posted 2023-09-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2023-10

CONDITIONS: Parkinson; Parkinson Disease; Parkinson's Disease and Parkinsonism
Keywords: Cyclops®; Levodopa Cyclops®; Cyclops; Inhaled levodopa; OFF episodes; motor fluctuations
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; cyclopia sequence | interventions — Dihydroxyphenylalanine

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, crossover, comparative bioavailability study in healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test 1 - Levodopa Cyclops® 45 mg (Experimental): 1 pre-filled single-use Levodopa Cyclops® (= 45 mg levodopa)
  Interventions: Combination Product: Levodopa Cyclops®
- Test 2 - Levodopa Cyclops® 90 mg (Experimental): 2 pre-filled single-use Levodopa Cyclops® devices (= 90 mg levodopa)
  Interventions: Combination Product: Levodopa Cyclops®
- Test 3 - Levodopa Cyclops™ 135 mg (Experimental): 3 pre-filled single-use Levodopa Cyclops® devices (= 135 mg levodopa)
  Interventions: Combination Product: Levodopa Cyclops®
- Reference - Inbrija® 84 mg (Active Comparator): 2 Inbrija® capsules (42 mg levodopa per capsule) from the Arcus® dry powder inhaler
  Interventions: Combination Product: INBRIJA®

INTERVENTIONS:
Combination Product: Levodopa Cyclops® — Orally inhaled dry powder levodopa from the Cyclops® dry powder inhaler
  Arms: Test 1 - Levodopa Cyclops® 45 mg; Test 2 - Levodopa Cyclops® 90 mg; Test 3 - Levodopa Cyclops™ 135 mg
Combination Product: INBRIJA® — Orally inhaled dry powder levodopa from the ARCUS® dry powder inhaler
  Arms: Reference - Inbrija® 84 mg

SUMMARY:
Patients with Parkinson's disease (PD) are commonly treated with a combination of levodopa and a decarboxylase inhibitor (DCI). However, many PD patients experience motor fluctuations (OFF episodes), even with their regular levodopa/DCI treatment.

This unmet medical need was addressed by the approval of INBRIJA®, an orally inhaled product, for producing therapeutic relief during the OFF episodes. INBRIJA® is a capsule-based inhaler system and in order to administer the full dose of levodopa, the patients need to inhale the contents of two capsules. In order to administer the full dose of levodopa, patients need to inhale the contents of two capsules. Since the INBRIJA® device is a standalone and reusable unit, the patients have to load the capsule prior to inhalation several times a day during the OFF episodes (except early-morning OFF) to get relief. Also, the INBRIJA® device is repeatedly used by PD patients and therefore needs to be properly cleaned to avoid contamination.

PureIMS is developing a more user-friendly alternative called Levodopa Cyclops®, a pre-filled drug-device combination of levodopa inhalation powder for use with the Cyclops® dry powder inhaler. Due to the nature of the Cyclops®, it offers PD patients greater ease and convenience in use. Moreover, the device's moderate to high resistance to airflow and minimal use of excipients suggests minimal cough episodes during oral inhalation.

The current study is planned in order to determine the dose at which comparative bioavailability of Levodopa Cyclops® will be reached compared to INBRIJA®.

DETAILED DESCRIPTION:
Patients with Parkinson's disease (PD) are commonly treated with a combination of levodopa and a decarboxylase inhibitor (DCI). However, many PD patients experience motor fluctuations (OFF episodes), even with their regular levodopa/DCI treatment. This unmet medical need was addressed by the approval of INBRIJA®, an orally inhaled product, which releases levodopa in the systemic circulation for producing therapeutic relief during the OFF episodes.

The INBRIJA® inhaler system is based on a spray-dried powder and contains 90% of levodopa, 8% dipalmitoyl phosphatidylcholine, and 2% sodium chloride. In order to administer the full dose of levodopa, patients need to inhale the contents of two capsules. Since the INBRIJA® device is a standalone and reusable unit, the patients have to load the capsule prior to inhalation several times a day during the OFF episodes (except early-morning OFF) to get relief. Also, the INBRIJA® device is repeatedly used by PD patients and therefore needs to be properly cleaned to avoid contamination.

PureIMS is developing a drug-device combination product called Levodopa Cyclops®, a pre-filled drug-device combination of levodopa inhalation powder for use with the Cyclops® dry powder inhaler. The ready-to-use Cyclops® carries a high load of drug (i.e., 98% levodopa with only 2% L-leucine serving as the excipient). Due to the nature of the Cyclops®, it offers PD patients greater ease and convenience in use. Moreover, the device's moderate to high resistance to airflow and minimal use of excipients suggests minimal cough episodes during oral inhalation.

Levodopa Cyclops® has shown safety and tolerability in PD patients with no reports of cough episodes. The pharmacokinetics (PK) at 30, 60 and 90 mg Levodopa Cyclops® doses show a dose proportional increase of exposure (Cmax and AUC) with a rapid attainment of Cmax (within 10 minutes after oral inhalation using Levodopa Cyclops®).

PureIMS plans to pursue drug development in the US via the 505(b)(2) regulatory pathway, referencing the safety and efficacy findings of the FDA for the approved levodopa inhaler INBRIJA®.

The current study is planned in order to determine the dose at which comparable relative bioavailability of Levodopa Cyclops® will be reached compared to INBRIJA®. The selected Levodopa Cyclops® dose will then be investigated against INBRIJA® in a formal comparative bioavailability study, in order to provide a PK bridge of Levodopa Cyclops® to the reference listed drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject
2. Age between 18 and 55 years (inclusive the date of signing informed consent)
3. Female subject who IS NOT of reproductive potential. A female subject who is NOT of reproductive potential is defined as one who:

   (i) has reached natural menopause (defined as at least 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone [FSH] levels in the postmenopausal range as determined by the local laboratory, or 12 months of spontaneous amenorrhea); (ii) is 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy; or (iii) has undergone bilateral tubal ligation. Spontaneous amenorrhea does not include cases for which there is an underlying disease that causes amenorrhea (e.g. anorexia nervosa)
4. Female subject who IS of reproductive potential and uses reliable contraception method and/or is willing to use adequate birth control methods starting from the time of consent through 30 days after the last dose of study therapy

   List of medically accepted contraceptive methods (used at least 4 weeks prior screening visit and not to be changed for the duration of the study):
   * Combination of a barrier method and spermicides (film, jelly, foam): e.g. female/ male condoms with spermicides, as well as diaphragm/ cervical cap/ contraceptive sponge with spermicides.
   * Hormonal methods: combined estrogen/progestin injectable and oral contraceptives; progestin injectable and oral contraceptives; implants (Nexplanon®), vaginal ring (NuvaRing®), skin patch (Xulane®) and contraceptive injection (Depo-Provera®).
   * Intrauterine devices (IUD): inert or copper IUD (ParaGard®), hormonal IUD (Mirena®, Skyla®, Kyleena®).
5. Physically and mentally healthy as judged by means of medical and standard laboratory examination
6. Non-smokers or ex-smokers (stopped at least 6 months ago) with a smoking history of ≤5 pack-year equivalents (1 pack-year equivalent is equal to smoking 1 pack per day for 1 year) and non-users of othernicotine containing products, confirmed by urine cotinine test
7. BMI within the range (including the borders) of 18.0 to 30.0 kg/m2
8. Normal spirometry values at screening (forced expiratory volume in one second [FEV1] and forced vital capacity [FVC] between 80% and 120% of the average value regarding age, height, gender and ethnicity (acc. to ECCS/ERS)1
9. Informed consent given in written form according to chapter 5.4 of clinical trial protocol

Exclusion Criteria:

1. Participation in another clinical trial at same time or within 90 days before screening visit (calculated from the date of the final examination of the previous study)
2. Randomization into the present trial more than once
3. Pregnant and/or nursing women. Positive pregnancy test
4. Weight of less than 40 kg
5. Blood donation or blood loss including plasmapheresis of >500 mL within 90 days before screening visit
6. History of drug abuse or use of illegal drugs: use of soft drugs, e.g. marihuana within 6 months before screening visit or hard drugs, e.g. cocaine, amphetamines, phencyclidine within 1 year before screening visit
7. Alcohol abuse, i.e. regular use of more than 2 units of alcohol per day or 10 units per week or a history of alcoholism (one unit of alcohol equals 250 mL beer, 125 mL wine or 25 mL spirits) or recovered alcoholics
8. Regular consumption of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine containing sodas, chocolate) equivalent to more than 500 mg methylxanthines per day
9. Positive drug screening
10. Positive alcohol test
11. History of significant multiple and/or severe allergies (including latex allergy, asthma or bronchial hyperreactivity), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
12. Any history of drug hypersensitivity (especially to the active ingredient levodopa of the Test and Reference IMPs and to the active ingredient carbidopa of the AxMP) or intolerance to any sugar (e.g. fructose, glucose, or lactose)
13. Presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, hematological, gastrointestinal, neurological, psychiatric or other diseases
14. Clinically significant illness within 4 weeks before screening visit
15. Major surgery of the gastrointestinal tract except for appendectomy
16. Any chronic disease which might interfere with resorption, distribution, metabolism or excretion of the drug
17. History of difficulty in swallowing
18. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies
19. Administration of depot injectable solutions or medications with a halflife >1 week (including study medications) within 6 months before screening visit
20. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before screening visit
21. Intake or administration of any systemic or topical medication (including OTC medication and especially intake of antacids e.g. aluminum hydroxide, magnesium hydroxide, and simethicone or herbal medication e.g. St. John's wort, kava kava) within 2 weeks before screening visit
22. Medication with drugs known to alter the major organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within 60 days before screening visit
23. Systolic blood pressure outside the range of 100 to 135 mmHg and/or diastolic blood pressure outside the range of 60 to 90 mmHg
24. Pulse rate outside the range of 50 to 90 beats/min
25. Respiratory rate outside the range of 12-16 breaths/min
26. Axillary body temperature outside the interval of 35.5 to 37.1°C
27. Any clinically significant abnormality of the resting ECG (12-lead)
28. Laboratory values outside normal range with clinical relevance
29. Special diet due to any reason, e.g. vegetarians
30. Subjects who are known or suspected:

    * not to comply with the study directives
    * not to be reliable or trustworthy
    * not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed
    * to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in
    * subject is in custody or submitted to an institution due to a judicial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
The dose at which comparative bioavailability of levodopa will be reached between Levodopa Cyclops® versus Inbrija® | 5 days
  The primary objective of the present trial is to determine the dose at which comparative bioavailability of levodopa will be reached between Levodopa Cyclops® versus Inbrija® in healthy adult subjects after an oral inhalation of a single dose of 45, 90 and 135 mg levodopa under fasting conditions administered with 50 mg carbidopa one hour prior IMP administration in 3 study periods and after a single dose of 66 mg levodopa delivered dose (2 hard capsules containing 42 mg levodopa each) of Inbrija® administered with carbidopa 50 mg one hour prior to IMP administration in a fourth study period.

SECONDARY OUTCOMES:
The time to reach a levodopa plasma concentration above 400 ng/mL as a measure for the onset of action. | 5 days
  In the scientific literature it is stated that levodopa is effective at plasma concentrations above 400 ng/mL, therefore, the time it takes to reach this concentration with Levodopa Cyclops® and Inbrija® is of interest and is indicative for the onset of action.
The time above a levodopa plasma concentration 400 ng/mL as a measure for the duration of effect. | 5 days
  In the scientific literature it is stated that levodopa is effective at plasma concentrations above 400 ng/mL, therefore, the time above this concentration after a Levodopa Cyclops® dose or Inbrija® dose is of interest.
Safety and tolerability of Levodopa Cyclops® by measuring vital signs, laboratory examination and adverse events questioning | 5 days
  Before and after the study:
  * Vital signs (body temperature, pulse rate, respiratory rate, blood pressure)
  * 12-lead ECG
  * Laboratory examination blood and urine (Hematology, Chemistry, Serology, Serum FSH in females, Urinalysis)
  After each dose:
  * Adverse event questioning
  * Vital signs (pulse rate and blood pressure) measurement at 50 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Bogdanov, MD, Principal Investigator — Bed space for short term stay at Diagnostic & Consultative Centre 'Ascendent' Ltd.
Locations (1):
- Bed space for short term stay at Diagnostic & Consultative Centre 'Ascendent' Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No